CLINICAL TRIAL: NCT00004418
Title: Study of Glyceryl Trierucate and Glyceryl Trioleate (Lorenzo's Oil) Therapy in Male Children With Adrenoleukodystrophy
Brief Title: Effect of Glycerol Trierucate on Clinical Course of Adrenoleukodystrophy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: No funding, move to expanded access
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 199/13312; Nutricia-Loma Linda (Other Grant/Funding Number: Nutricia-Loma Linda); KKI-FDR000685 (Other: FDA)
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Results first posted 2020-10-23 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Adrenoleukodystrophy
Keywords: adrenoleukodystrophy; inborn errors of metabolism; rare disease; sphingolipidoses
MeSH Terms: conditions — Adrenoleukodystrophy; Metabolism, Inborn Errors; Rare Diseases; Sphingolipidoses | interventions — trierucate; Triolein; Lorenzo's oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Glyceryl trierucate/glyceryl trioleate (Experimental): Treatment of all enrolled participants. Dosage form is a liquid oil taken orally. Dose is to provide 20% of daily calories. Daily for duration of trial
  Interventions: Drug: glyceryl trierucate/glyceryl trioleate

INTERVENTIONS:
Drug: glyceryl trierucate/glyceryl trioleate — Administration of glyceryl trierucate/glyceryl trioleate
  Other Names: Lorenzo's oil

SUMMARY:
OBJECTIVES: I. Evaluate the clinical efficacy of combination glyceryl trierucate and glyceryl trioleate (Lorenzo's Oil) therapy in boys with X-linked adrenoleukodystrophy.

II. Compare the frequency and severity of neurological disability of study patients with untreated historical controls.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is an open label study. Patients must follow dietary instructions as provided by the investigator. Patients receive 2-4 tablespoons of a mixture of glyceryl trierucate and glyceryl trioleate oil once daily. Patients complete a neuropsychological scoring scale questionnaire to measure neurological disability. Patients undergo physical examinations including magnetic resonance imaging and magnetic resonance spectroscopy of the head.

Patients are followed monthly for 6 months, then every 3 months until they reach the age of 13 years or death.

ELIGIBILITY:
Inclusion criteria.

1. Boys between the age of 18 months and 8 years of age
2. Biochemically proven asymptomatic X-linked adrenoleukodystrophy determined by elevation of very long chain fatty acids or DNA analysis.
3. Platelet count in normal range

Exclusion criteria.

1. Abnormal MRI consistent with childhood cerebral disease
2. Boys who have undergone bone marrow transplantation
3. Other medical condition which in the opinion of the investigator prevents evaluation or treatment

Ages: 18 Months to 8 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — males only
Enrollment: 126 (Actual)
Dates: Start 1998-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerald V Raymond, M.D., Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (2):
- United States (2):
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: An open trial of Lorenzo's oil spanning decades (1998-2013). Centered at the Kennedy Krieger.
Groups:
- GTO/GTE Treatment: Intervention: A mixture of glycerol trierucate (GTE) in glycerol trioleate (GTO) in combination with a diet low in saturated fats.
  GTO/GTE orally; 30-60 ml daily for study period
  glyceryl trierucate: Glyceryl trierucate is an oil to reduce very long chain fatty acids
  glyceryl trioleate: Patients receive 2-4 tablespoons of a mixture of glyceryl trierucate and glyceryl trioleate oil once daily.
Period: Overall Study
Arm/Group | GTO/GTE Treatment
Started | 126
Completed | 126 (The definition of completed is until the subject wished to stop taking the oil.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | GTO/GTE Treatment
Number analyzed (Participants) | 126
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 126
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 3.25 [1.5 to 8]
Sex: Female, Male [Count of Participants; unit: Participants] — Male children only were eligible for this study.
  Participants
    Female | 0
    Male | 126
Region of Enrollment [Number; unit: participants]
  United States | 126

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Very Long Chain Fatty Acids (VLCFA) Blood Levels
Description: we will assess the change in very long-chain fatty acids as determined by reduction of blood level baseline C26:0 level.
Time Frame: Baseline, an average of 10 years, up to age 13
Measure: Mean (Full Range); unit: mcg/mL
Arm/Group | GTO/GTE Treatment
Number analyzed (Participants) | 126
mcg/mL | 0.41 [0.05 to 0.41]

2. Secondary Outcome: Number of Participants With T2 MRI Abnormality
Description: We used MRI to determine the number of participants with T2 MRI abnormality indicating childhood Adrenoleukodystrophy (ALD).
Time Frame: 10 years
Measure: Count of Participants; unit: Participants
Arm/Group | GTO/GTE Treatment
Number analyzed (Participants) | 126
Participants | 0

ADVERSE EVENTS:
Time Frame: 10 years (throughout the study)
Arm/Group | GTO/GTE Treatment
All-Cause Mortality (participants affected / at risk) | 1/126
Serious Adverse Events (participants affected / at risk) | 3/126
Other Adverse Events (participants affected / at risk) | 1/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GTO/GTE Treatment (N=126)
Death (Endocrine disorders) | 1 (1) — Subject had profound adrenal crisis and died
adrenal crisis (Endocrine disorders) | 2 (2) — Two events of adrenal crisis
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GTO/GTE Treatment (N=126)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) — Low platelet count defined as <80, 000
Elevation in liver function tests (Hepatobiliary disorders) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes